CLINICAL TRIAL: NCT01392638
Title: Influence of the Nitric Oxide Synthase T-786C Polymorphism on the Response to Acute Inhibition of Phosphodiesterase 5 in Resistant Hypertension
Brief Title: Effects of Sildenafil in Resistant Hypertensives and Genetic Polymorphism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Heitor Moreno Junior, MD. PhD, University of Campinas, Brazil
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE-0758.0.146.000-09; FAPESP (Other: 2009/13774-9)
Record Dates: First submitted 2011-01-25; First posted 2011-07-12 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Hypertension
Keywords: Sildenafil; Nitric oxide synthase; Polymorphism; Hemodynamics
MeSH Terms: conditions — Hypertension | interventions — Sugars; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- sugar pill (Placebo Comparator): Intervention: sugar pill
  Interventions: Other: sugar pill
- sildenafil (Active Comparator): Intervention: sildenafil citrate
  Interventions: Drug: sildenafil

INTERVENTIONS:
Other: sugar pill — Sugar pills: 37.5, 50.0, and 100.0 mg each 30 minutes.
  Other Names: No brand name.
  Arms: sugar pill
Drug: sildenafil — Sildenafil pills: 37.5, 50.0, and 100.0 mg each 30 minutes.
  Other Names: Viagra, Pfizzer Lab., USA
  Arms: sildenafil

SUMMARY:
Sildenafil citrate slightly reduces blood pressure in treated hypertensives patients. However, it is unknown if the simultaneous use of sildenafil plus, at least, 3 classes of antihypertensive agents in patients with resistant arterial hypertension may have a synergic effect on the patients blood pressure. Moreover, sildenafil improves the endogen nitric oxide effects. The nitric oxide is an important signaling molecule in the body that contributes to vessel homeostasis by inhibiting vascular smooth muscle contraction and growth. Hypertension often impaired NO pathways. Nitric oxide is produced by an enzyme, called nitric oxide synthase (NOS3), that show some genetics variants, which means that this enzyme can be different from person to person. Therefore, the objective of the present study is to examine the influence of a genetic variant (known to affect NOS3 levels) in sildenafil acute effects on hemodynamic and cardiovascular function. The investigators hypothesis is that individuals with the genetic variant associated to higher levels of NOS3 will have more benefits from sildenafil treatment.

DETAILED DESCRIPTION:
Endothelial dysfunction is one of the mechanisms involved in the maintenance of the high blood pressure levels in resistants hypertensives patients, which is directly related to the NO-GMPc pathway. The phosphodiesterase 5 inhibitor, sildenafil citrate, slightly reduces systolic and diastolic blood pressures in treated hypertensives patients. However, it is unknown if the simultaneous use of sildenafil plus, at least, 3 classes of antihypertensive agents in patients with resistant arterial hypertension may have a synergic effect on the patients blood pressure. Moreover, sildenafil improves the endogen nitric oxide effects produced by eNOS. Therefore, since the genetics polymorphisms of eNOS can affect the NO tissue levels, it seems reasonable to suppose that the acute effects of sildenafil may be modulated by them. Objective: To examine the influence of the T-786C polymorphism of eNOS gene in sildenafil acute effects on hemodynamic and cardiovascular function in resistant hypertensives patients. Casuistics and Methods: Around 120 patients with HAR will be genotyped for the T-786C eNOS polymorphism, from which the investigators will enroll in this study 15 patients with TT genotype and 15 patients with CC genotype. The patients will be monitored with the Portapres system (non-invasive hemodynamic). After basal records of the studied variables, increasing doses of sildenafil will be administrated (37.5, 50.0 e 100.0 mg). Five minutes before each new dose, the studied variables will be recorded again. Hypothesis: The investigators hypothesize that the sildenafil, besides the anti-ischemic effect, will improve the patients hemodynamic status and, moreover, that it will occur a modulation of this effect by the T-786C polymorphism.

ELIGIBILITY:
Inclusion Criteria:

* resistant hypertensive (according to Resistant Hypertension - AHA Statement - 2008);
* compliance with antihypertensive treatment;
* age >35 years;
* diastolic dysfunction

Exclusion Criteria:

* valvulopathy
* decompensated heart failure
* important cardiac arrhythmias
* nephropathy
* hepatopathy
* autoimmune disease
* tabagism
* decompensated diabetes
* uncontrolled dislipidemia

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Cardiac Output, total peripheral resistance, mean arterial pressure | Each 30 minutes
  Hemodynamic measures each 30 minutes

SECONDARY OUTCOMES:
Left ventricular diastolic function parameters, endothelial function | Pre- and post-sildenafil accumulated doses
  Assessment of how hemodynamic changes determined by sildenafil would affect endothelial and left ventricular diastolic parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Heitor Moreno, PhD, Principal Investigator — Faculty of Medical Sciences - Unicamp
Locations (1):
- Laboratory of Cardiovascular Pharmacology - FCM - Unicamp, Campinas, São Paulo, Brazil